CLINICAL TRIAL: NCT06767657
Title: Multicenter, Open-label Randomized Study Comparing Urgent Carotid Endarterectomy (CEA) (within 72 Hours) Versus Delayed CEA (after 72 Hours) in Patients with Symptomatic Carotid Stenosis (SPREAD-STACI II)
Brief Title: Urgent Carotid Endarterectomy (CEA) Versus Delayed CEA in Symptomatic Carotid Stenosis (SPREAD-STACI II)
Acronym: Time_to_sCEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Italian Society of Vascular and Endovascular Surgery (Other)
Responsible Party: Principal Investigator, EMILIANO CHISCI, Principal Investigator, Head of Endovascular Aortic UNIT, San Giovanni di Dio Hospital, USL Toscana Centro, Florence, ITALY, Italian Society of Vascular and Endovascular Surgery
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SPREAD STACI TRIAL II
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Ischemic; Transient Ischemic Accident; Endarterectomy, Carotid; Stroke Prevention
Keywords: stroke; endarterectomy; transient ischemic accident; stroke prevention
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: The study will evaluate the same surgical procedure, carotid endarterectomy (CEA), which involves the removal of the atherosclerotic plaque causing thromboembolism or hemodynamically significant stenosis. This will be performed in two different timeframes:
  Within 72 hours of the ischemic symptom. Between 72 hours and 14 days after the symptom.
  The two study groups will not differ in the type of treatment offered but only in the timing of its execution.
  No experimental procedures will be conducted. Whether CEA is performed within 72 hours or after this period, the surgical procedure will adhere fully to the current guidelines.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : Within 72 hours of the ischemic symptom (Experimental): The study will evaluate the same surgical procedure, carotid endarterectomy (CEA), which involves the removal of the atherosclerotic plaque causing thromboembolism or hemodynamically significant stenosis. This will be performed in two different timeframes:
  GROUP A : Within 72 hours of the ischemic symptom. GROUP B: Between 72 hours and 14 days after the symptom.
  The two study groups will not differ in the type of treatment offered but only in the timing of its execution.
  No experimental procedures will be conducted. Whether CEA is performed within 72 hours or after this period, the surgical procedure will adhere fully to the current guidelines.
  Interventions: Procedure: CEA (carotid endarterectomy)
- Group B: Between 72 hours and 14 days after the ischemic symptom (Active Comparator): see above
  Interventions: Procedure: CEA (carotid endarterectomy)

INTERVENTIONS:
Procedure: CEA (carotid endarterectomy) — Intervention (CEA) is associated to both arms (group A and B)

SUMMARY:
In patients with internal carotid artery (ICA) stenosis of 50% or greater (measured according to the criteria of the North American Symptomatic Carotid Endarterectomy Trial (NASCET)) who have experienced a transient ischemic attack (TIA) or minor ipsilateral stroke, carotid endarterectomy (CEA) offers maximum benefit if performed within 15 days of the initial ischemic symptom. National and international guidelines recommend surgical treatment (CEA) within this timeframe; however, no studies have specifically evaluated the optimal timing for CEA after a TIA or minor stroke.

It is well established that the risk of a major stroke is highest in the first few days following a transient ischemic attack or minor stroke and then decreases over the subsequent days and weeks.

This raises the hypothesis that performing an urgent carotid endarterectomy (within 3 days) may provide greater benefit compared to a delayed procedure (between 4 and 15 days).

DETAILED DESCRIPTION:
Background and Rationale

In patients with internal carotid artery (ICA) stenosis of 50% or greater (measured according to the criteria of the North American Symptomatic Carotid Endarterectomy Trial (NASCET)) who have experienced a transient ischemic attack (TIA) or minor ipsilateral stroke, carotid endarterectomy (CEA) offers maximum benefit if performed within 15 days of the initial ischemic symptom. National and international guidelines recommend surgical treatment (CEA) within this timeframe; however, no studies have specifically evaluated the optimal timing for CEA after TIA or minor stroke.

It is well established that the risk of a major stroke is highest in the first few days following a transient ischemic attack or minor stroke and then decreases over the subsequent days and weeks. This raises the hypothesis that performing an urgent carotid endarterectomy (within 3 days) may provide greater benefit compared to a delayed procedure (between 4 and 15 days).

Study Objectives

Primary Endpoint

To demonstrate that CEA for symptomatic ICA stenosis of 50% or greater (NASCET criteria) performed urgently within 72 hours of the onset of the ischemic symptom (TIA or minor stroke) is more effective than delayed CEA (performed after 72 hours but within 15 days) in reducing the risk of death, any type of stroke, and myocardial infarction within 90 days of the ischemic event.

Secondary Endpoints

To demonstrate that urgent CEA (within 72 hours of symptom onset) is more effective than delayed CEA (after 72 hours but within 15 days) in reducing the risk of ipsilateral ischemic stroke within 90 days of the ischemic event.

To identify potential subgroups of patients who benefit more from urgent CEA compared to delayed CEA.

To demonstrate that urgent CEA (within 72 hours) is as safe as delayed CEA (after 72 hours) in terms of the risk of cerebral hemorrhagic complications.

Study Design

This is a prospective, randomized, multicenter, controlled, non-profit interventional study with blinded follow-up at 90 days by the neurologist/internist investigator. The study is coordinated by the Vascular Surgery Unit (UOC) at San Giovanni di Dio Hospital, USL TOSCANA CENTRO, in collaboration with the Vascular Surgery Units listed above. All patients treated at the participating centers are eligible for inclusion if they meet the inclusion and exclusion criteria and provide informed consent to participate in the study.

The study does not introduce modifications or conflicts with standard clinical practice, as all enrolled and randomized patients (whether within or after 72 hours) will undergo surgical treatment (CEA) within 15 days of the index symptom, in accordance with national and international guidelines.

Study Population

Number of patients to be enrolled: 456

Withdrawal Criteria Patients may withdraw from the study at any time.

Interventions

The study will evaluate the same surgical procedure, carotid endarterectomy (CEA), which involves the removal of the atherosclerotic plaque causing thromboembolism or hemodynamically significant stenosis. This will be performed in two different timeframes:

Within 72 hours of the ischemic symptom. Between 72 hours and 14 days after the symptom.

The two study groups will not differ in the type of treatment offered but only in the timing of its execution.

No experimental procedures will be conducted. Whether CEA is performed within 72 hours or after this period, the surgical procedure will adhere fully to the current guidelines.

Assessment of Potential Benefit/Risk for the Study Population

The morbidity and mortality risk for the study participants is expected to be within the 6% limit for stroke/mortality at 30 days, as defined by the safety threshold in the literature and by national and international guidelines.

If this threshold (stroke/mortality at 30 days ≥ 6%) is exceeded in either group, the study will be terminated for safety reasons.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Patients presenting with the following characteristics:

De novo stenosis of the carotid bifurcation and/or internal carotid artery origin, equal to or greater than 50% (NASCET method), diagnosed by color Doppler ultrasound, MR angiography (MRA), CT angiography (CTA), or catheter angiography.

TIA or minor ischemic stroke (NIHSS ≤ 5) ipsilateral to the carotid stenosis, occurring within the previous 24 hours.

Preserved consciousness and neurologically stable symptoms. No evidence of ongoing cerebral ischemia, or evidence of cerebral ischemia with a diameter <25 mm.

Age between 45 and 90 years. ASA score < 4. Ability to comply with follow-up requirements as specified. Willingness to provide informed consent for participation in the study.

A patient with an NIHSS ≤ 5 who is aphasic may be unable to provide consent. In these cases:

The attending physician assesses the feasibility of including the patient. Family members are informed but, under Italian law, cannot provide consent. A third-party physician certifies that the patient meets the inclusion criteria.

The attending physician signs the appropriate form, and randomization proceeds. If and when the patient regains the ability to provide or refuse consent, the informed consent form will be presented to them. Should they decline, their data will be removed from the study database.

Additionally, the study includes patients who underwent thrombolysis and/or mechanical thrombectomy after the onset of the index symptom, followed by a brain CT/MRI without secondary cerebral hemorrhage (PH1, PH2, or PHr).

Exclusion Criteria:

Stenosis < 50% (NASCET method) at the bifurcation and/or internal carotid artery origin, diagnosed by ECD, CTA, or MRA.

Carotid thrombosis or dissection. NIHSS > 5. Cerebral hemorrhage. Impaired consciousness or neurologically unstable condition. Cancer, any condition with a poor prognosis, major cardiopathy, or any severe neurological disorder.

CT or MRI evidence of cerebral ischemia > 25 mm in diameter. CT or MRI evidence of cerebral lesions of uncertain origin. Recurrent TIA or stroke-in-evolution. Age < 45 years or > 90 years. ASA risk score = 4. Lack of informed consent. Inability to undergo CEA within 72 hours of the initial ischemic symptom. Inability to participate in a 90-day follow-up after the initial ischemic symptom.

Previous CEA or stenting of the examined carotid artery.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related death, any type of stroke, and myocardial infarction events as assessed by CTCAE v4.0 | From enrollment to 90 days follow-up from CEA
  Number of patients experiencing death, any type of stroke, and myocardial infarction within 90 days of the ischemic event in group A and B (numerical values)

SECONDARY OUTCOMES:
Number of participants with treatment-related ipsilateral ischemic stroke events as assessed by CTCAE v4.0 | From enrollment to 90 days follow-up from CEA
  Number of patients experiencing ipsilateral ischemic stroke within 90 days of the ischemic event in group A and B. (numerical values)
Number of participants with treatment-related cerebral hemorrhagic events as assessed by CTCAE v4.0 | From enrollment to 90 days follow-up from CEA
  To demonstrate that urgent CEA (within 72 hours) is as safe as delayed CEA (after 72 hours) in terms of number of cerebral hemorrhagic events.

CONTACTS AND LOCATIONS:
Locations (1):
- Usl Toscana Centro, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified Participant-Level Data: Informed consent templates , CRF Baseline clinical characteristics, including NIHSS score, comorbidities, and ASA score.) Diagnostic results related to carotid stenosis.Treatment details, including timing of CEA (urgent vs. delayed) and any perioperative interventions.
  Outcomes data, including: Incidence of stroke (all types), myocardial infarction, and death within 30 and 90 days.Neurological complications (e.g., ipsilateral ischemic stroke). Safety endpoints, including complications such as hemorrhagic stroke and other adverse events.
  Detailed study protocol outlining eligibility criteria, interventions, and endpoints. Statistical analysis plans used to to evaluate primary and secondary endpoints.
  Access will be granted after completion of the study and publication of the primary results.Requests must include a proposal for a secondary analysis, a data-sharing agreement, and a commitment to maintaining data confidentiality
Supporting Information: Study Protocol, CSR
Time Frame: form January 2025 to December 2028
Access Criteria: The IPD (Individual Participant Data) can be accessed by all members of the Italian Society of Vascular and Endovascular Surgery (SICVE) who submit a direct access request via the SICVE web address at https://www.anughea.ai/wp-login.php.
URL: https://www.anughea.ai/

REFERENCES:
- [Background] Naylor AR. Occam's razor: Intervene early to prevent more strokes! J Vasc Surg. 2008 Oct;48(4):1053-9. doi: 10.1016/j.jvs.2008.06.044. Epub 2008 Aug 23. PMID 18723309
- [Background] Nordanstig A, Rosengren L, Stromberg S, Osterberg K, Karlsson L, Bergstrom G, Fekete Z, Jood K. Editor's Choice - Very Urgent Carotid Endarterectomy is Associated with an Increased Procedural Risk: The Carotid Alarm Study. Eur J Vasc Endovasc Surg. 2017 Sep;54(3):278-286. doi: 10.1016/j.ejvs.2017.06.017. Epub 2017 Jul 26. PMID 28755855
- [Background] Kakkos SK, Vega de Ceniga M, Naylor R. A Systematic Review and Meta-analysis of Peri-Procedural Outcomes in Patients Undergoing Carotid Interventions Following Thrombolysis. Eur J Vasc Endovasc Surg. 2021 Sep;62(3):340-349. doi: 10.1016/j.ejvs.2021.06.003. Epub 2021 Jul 12. PMID 34266765
- [Background] Coelho A, Peixoto J, Mansilha A, Naylor AR, de Borst GJ. Editor's Choice - Timing of Carotid Intervention in Symptomatic Carotid Artery Stenosis: A Systematic Review and Meta-Analysis. Eur J Vasc Endovasc Surg. 2022 Jan;63(1):3-23. doi: 10.1016/j.ejvs.2021.08.021. Epub 2021 Dec 23. PMID 34953681
- [Background] Stromberg S, Gelin J, Osterberg T, Bergstrom GM, Karlstrom L, Osterberg K; Swedish Vascular Registry (Swedvasc) Steering Committee. Very urgent carotid endarterectomy confers increased procedural risk. Stroke. 2012 May;43(5):1331-5. doi: 10.1161/STROKEAHA.111.639344. Epub 2012 Mar 15. PMID 22426315
- [Background] Loftus IM, Paraskevas KI, Johal A, Waton S, Heikkila K, Naylor AR, Cromwell DA. Editor's Choice - Delays to Surgery and Procedural Risks Following Carotid Endarterectomy in the UK National Vascular Registry. Eur J Vasc Endovasc Surg. 2016 Oct;52(4):438-443. doi: 10.1016/j.ejvs.2016.05.031. Epub 2016 Jun 28. PMID 27364857
- [Background] Naylor R, Rantner B, Ancetti S, de Borst GJ, De Carlo M, Halliday A, Kakkos SK, Markus HS, McCabe DJH, Sillesen H, van den Berg JC, Vega de Ceniga M, Venermo MA, Vermassen FEG, Esvs Guidelines Committee, Antoniou GA, Bastos Goncalves F, Bjorck M, Chakfe N, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kolh P, Koncar IB, Lindholt JS, Mees BME, Resch TA, Trimarchi S, Tulamo R, Twine CP, Wanhainen A, Document Reviewers, Bellmunt-Montoya S, Bulbulia R, Darling RC 3rd, Eckstein HH, Giannoukas A, Koelemay MJW, Lindstrom D, Schermerhorn M, Stone DH. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on the Management of Atherosclerotic Carotid and Vertebral Artery Disease. Eur J Vasc Endovasc Surg. 2023 Jan;65(1):7-111. doi: 10.1016/j.ejvs.2022.04.011. Epub 2022 May 20. No abstract available. PMID 35598721
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Lanza G, Orso M, Alba G, Bevilacqua S, Capoccia L, Cappelli A, Carrafiello G, Cernetti C, Diomedi M, Dorigo W, Faggioli G, Giannace V, Giannandrea D, Giannetta M, Lanza J, Lessiani G, Marone EM, Mazzaccaro D, Migliacci R, Nano G, Pagliariccio G, Petruzzellis M, Plutino A, Pomatto S, Pulli R, Reale N, Santalucia P, Sirignano P, Ticozzelli G, Vacirca A, Visco E. Guideline on carotid surgery for stroke prevention: updates from the Italian Society of Vascular and Endovascular Surgery. A trend towards personalized medicine. J Cardiovasc Surg (Torino). 2022 Aug;63(4):471-491. doi: 10.23736/S0021-9509.22.12368-2. PMID 35848869
- [Background] Lanza G, Ricci S, Speziale F, Toni D, Sbarigia E, Setacci C, Pratesi C, Somalvico F, Zaninelli A, Gensini GF. SPREAD-STACI study: a protocol for a randomized multicenter clinical trial comparing urgent with delayed endarterectomy in symptomatic carotid artery stenosis. Int J Stroke. 2012 Jan;7(1):81-5. doi: 10.1111/j.1747-4949.2011.00699.x. Epub 2011 Dec 8. PMID 22151469